CLINICAL TRIAL: NCT05054998
Title: A Pilot Study of Dual Time Point FDG PET MR Imaging Optimization for the Evaluation of Brain Metastasis
Brief Title: Dual Time Point FDG PET/MRI Scan in Improving the Imaging Cancer Patients With Brain Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0435; NCI-2019-02459 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0435 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-09; First posted 2021-09-23 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (fludeoxyglucose F-18, PET/MRI) (Experimental): Patients receive fludeoxyglucose F-18 IV over approximately 1 minute and undergo a PET/MRI scan over 70 minutes. Within 5 hours of receiving fludeoxyglucose F-18, patients undergo a repeat PET/MRI scan over 30 minutes. Scans take place within 2 weeks before scheduled surgery and within 4-6 weeks after radiation treatment.
  Interventions: Radiation: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Radiation: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase IV trial studies how well delaying positron emission tomography (PET)/magnetic resonance imaging (MRI) scan after injection of fluorodeoxyglucose (FDG) can improve the imaging of patients with cancer that has spread to brain (brain metastases). FDG is a type of imaging agent that doctors use to help "see" the images on a scan more clearly. Delaying PET/MRI scan after injecting FDG may improve how well doctors can tell the difference between healthy and unhealthy tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the optimal fludeoxyglucose F-18 (fluorodeoxyglucose) positron emission tomography (FDG PET) imaging time post radiotracer administration that maximizes separation of activity between lesion and non-lesional parenchyma (measured as lesion/background [L/B] ratio) in patients with brain metastasis.

SECONDARY OBJECTIVE:

I. To identify genotypic factors in FDG tumor metabolism derived from metrics, including maximum standard uptake value (SUVmax), mean standard uptake value (SUVmean), total lesion glycolysis (TLG), mean tumor volume (MTV), and L/B ratio.

EXPLORATORY OBJECTIVES:

I. To identify patterns of metabolism derived from metrics, such as SUVmax, SUVmean, TLG, MTV, and L/B ratio, and magnetic resonance imaging metrics, such as regional perfusion abnormalities, apparent diffusion coefficient values, fractional diffusivity measures, and magnetic resonance spectroscopic finding.

II. To identify if post treatment changes in lesion metabolism from baseline correlate with treatment success.

OUTLINE:

Patients receive fludeoxyglucose F-18 intravenously (IV) over approximately 1 minute and undergo a PET/MRI scan over 70 minutes. Within 5 hours of receiving fludeoxyglucose F-18, patients undergo a repeat PET/MRI scan over 30 minutes. Scans take place within 2 weeks before scheduled surgery and within 4-6 weeks after radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pre-treatment adult patients with any solid organ metastasis and at least three intraaxial brain metastases including at least one enhancing > 10 mm lesion
* Rim or solid enhancing lesion(s) WITH a history of non-central nervous system (CNS) pathologic proven metastatic disease will be considered as a consensus between the referring radiation oncologist or neurosurgeon and a neuroradiology
* Planned surgery or radiation to the metastases
* Ability to undergo PET magnetic resonance (MR) examination

Exclusion Criteria:

* Known allergy to FDG or gadolinium based contrast agents
* History of impaired renal function (glomerular filtration rate [GFR] < 30)
* Pregnant women are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
assess the optimal fludeoxyglucose F-18 (fluorodeoxyglucose) positron emission tomography (FDG PET) imaging time post radiotracer administration that maximizes separation of activity between lesion and non-lesional parenchyma | through study completion, an average of a year

CONTACTS AND LOCATIONS:
Overall Officials: Dawid Schellingerhout, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org